CLINICAL TRIAL: NCT02621827
Title: Vitamin D Half-life in Pregnancy and Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Kerry Jones, Investigator scientist, Medical Research Council
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MRC SCC1229
Record Dates: First submitted 2015-11-27; First posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Pregnancy; Lactation
Keywords: vitamin D; Africa
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-pregnant, non-lactating (NPNL) (Experimental): NPNL women are age and parity matched to pregnant women. Each NPNL women is studied twice, approximately 3 months apart.
  At each study period the participant receives (as the intervention) a single oral dose of stable isotope labeled 25(OH)D3.
  Interventions: Other: Oral dose of stable isotope labeled 25(OH)D3
- Pregnant/Lactating (Experimental): Pregnant women receive (as the intervention) a single oral dose of stable isotope labeled 25(OH)D3. The same women are followed-up in lactation to repeat the same protocol.
  Interventions: Other: Oral dose of stable isotope labeled 25(OH)D3

INTERVENTIONS:
Other: Oral dose of stable isotope labeled 25(OH)D3 — At each measurement, women are given an oral dose of stable isotope labelled 25(OH)D3. Blood and urine samples are collected at baseline and on day 21 post-dose. Additional blood samples are collected post-dose on days 6,9,24,27 and 30.

SUMMARY:
This study measures the plasma half-life of 25-hydroxyvitamin D3 (25(OH)D3) in non-pregnant-non-lactating women, pregnant women at 30 wk gestational age and at 3 months post-partum in women who are exclusively breast-feeding.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Currently resident in West Kiang and planning to stay for the next 5 months
* Aged between 18 and 45 y

Pregnancy:

* > 20 wk < 30 wk pregnant (gestational age assessment by ultrasound)
* Singleton fetus

Lactation:

* Breast feeding

Exclusion Criteria:

All participants:

* Severe anaemia (haemoglobin < 7 g/dL) (as per ENID protocol)
* Known sickle cell anaemia
* Known to be asthmatic or allergic to peanuts (already excluded from ENID)
* Known history of liver, kidney, gut or malabsorption problems
* Other chronic condition
* On prescription medication
* Taking vitamin D supplements (> 200 IU/d)
* Broken bone in last 3 y
* Recent infection or illness (2 weeks prior to the start of a study period)
* Reported onset of menopause (already excluded from ENID)
* Malaria parasitemia (prior to study period)
* Unable to consent

Pregnant:

* Pregnancy-related complications or on discretion of mid-wife
* Known HIV positive

Lactation:

* Health problem of mother or infant that may affect feeding practices

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of stable isotope labeled 25(OH)D3 | Samples collected on day 6, 9, 21, 24, 27 and 30 post-dose
  The plasma half-life of 25(OH)D3 is calculated from the slope (k) of the disappearance of the stable isotope labeled 25(OH)D3 against time using the equation half-life=0.693/k

SECONDARY OUTCOMES:
Plasma concentration of vitamin D metabolites and related calciotropic hormones | Fasting plasma samples collected at baseline and 21 days post-dose
  Analytes: 25(OH)D3, 24,25(OH)2D3, 1,25(OH)2D, vitamin D binding protein, parathyroid hormone, albumin, ionised calcium, phosphate
Urinary concentration of calcium, phosphate, creatinine and cyclic adenosine monophosphate (cAMP) | Samples collected at baseline and 21 days post-dose
  2-hour fasting urine collection
Weighed dietary intake | 2 days within 30 days of dose
  Dietary nutrient intakes assessed by 2-day weighed food diary and nutrient intakes calculated using DINO (diet in nutrients out) analysis programme (Fitt et al, 2015)